CLINICAL TRIAL: NCT03105180
Title: The Effect of a Mixture of 2.7% Sorbitol-0.54% Mannitol Solution on Blood Coagulation: In-vitro, Observational Healthy-volunteer Study Using Rotational Thromboelastometry (ROTEM®)
Brief Title: Irrigating Fluid and Blood Coagulation
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Associate Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1703/386-303
Record Dates: First submitted 2017-03-29; First posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Blood Coagulation Disorder
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 0% dilution: Blood specimen which was diluted with 0% level using a mixture of 2.7% sorbitol-0.54% mannitol solution
- 10% dilution: Blood specimen which was diluted with 10% level using a mixture of 2.7% sorbitol-0.54% mannitol solution
  Interventions: Other: A mixture of 2.7% sorbitol-0.54% mannitol solution
- 20% dilution: Blood specimen which was diluted with 20% level using a mixture of 2.7% sorbitol-0.54% mannitol solution
  Interventions: Other: A mixture of 2.7% sorbitol-0.54% mannitol solution
- 40% dilution: Blood specimen which was diluted with 40% level using a mixture of 2.7% sorbitol-0.54% mannitol solution
  Interventions: Other: A mixture of 2.7% sorbitol-0.54% mannitol solution

INTERVENTIONS:
Other: A mixture of 2.7% sorbitol-0.54% mannitol solution — Venous blood was taken from 12 healthy volunteers and divided into four specimen bottles, which were diluted with different levels (0%, 10%, 20%, and 40%) using a mixture of 2.7% sorbitol-0.54% mannitol solution.
  Groups: 10% dilution; 20% dilution; 40% dilution

SUMMARY:
Irrigating fluid absorbed during the endoscopic surgery may alter whole blood coagulation. However, little is known about the dose-response relationships of hemodilution. The investigators have therefore performed the present study to measure the effect of a mixture of 2.7% sorbitol-0.54% mannitol solution on the coagulation pathway according to the hemodilution level using a rotational thromboelastometry (ROTEM®) tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* age: 20 to 65 years
* Body weight > 50 kg
* Volunteers who provided informed consent

Exclusion Criteria:

* Hematologic disease
* Anticoagulant medication

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
FIBTEM | during the rotational thromboelastometry analysis/ an average of 1 hour
  Fibrinolytic pathway values of rotational thromboelastometry analysis/ FIBTEM is s a proper noun which means the status of fibrinolytic coagulation pathway.

SECONDARY OUTCOMES:
INTEM | during the rotational thromboelastometry analysis/ an average of 1 hour
  Intrinsic pathway values of rotational thromboelastometry analysis/ INTEM is a proper noun which means the status of intrinsic coagulation pathway.
EXTEM | during the rotational thromboelastometry analysis/ an average of 1 hour
  Extrinsic pathway values of rotational thromboelastometry analysis/ EXTEM is a proper noun which means the status of extrinsic coagulation pathway.

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Seok Na, PhD, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No